CLINICAL TRIAL: NCT02633865
Title: Patient Participation in Free Cataract Surgery: The Low-income Elderly in Urban China
Brief Title: Patient Participation in Free Cataract Surgery
Status: Completed | Type: Observational
Sponsor: Sun Yat-sen University (Other)
Collaborators: Ministry of Health, China (Other Government)
Responsible Party: Principal Investigator, Haotian Lin, Principal Investigator, Home for Cataract Children, Zhongshan Ophthalmic Center, Sun Yat-sen University
Other Study IDs: CCPMOH2010-China11
Record Dates: First submitted 2015-12-09; First posted 2015-12-17 (Estimated); Last update posted 2016-04-20 (Estimated); Status verified 2016-04

CONDITIONS: Cataract
Keywords: patient characteristics
MeSH Terms: conditions — Cataract

STUDY DESIGN:
Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 9 Months
Oversight: Data Monitoring Committee: Yes

SUMMARY:
Age-related cataracts remain the leading cause of treatable blindness in China. The prevalence of cataract blindness continues to climb due to the expanding elderly subpopulation. Surgery is the only available treatment; however, the cataract surgical rate (CSR) in China remains relatively low relative to affluent countries or certain developing areas. Studies have reported that the primary barrier to cataract surgery is financial difficulty, and this challenge could be efficiently addressed by reducing the surgical fee or providing free cataract surgery. However, the prices, availability and affordability of medicines or medical services to the poor in China require further improvement. Although a host of free cataract screening and surgery programs have been widely implemented in rural areas of China, free cataract surgery programs have rarely been implemented in financially-challenged urban China. Even in Guangzhou, one of the largest metropolises in China, many low-income cataract patients, a neglected cohort, continue to need cataract surgery. A program titled "care for your eyes, lighten your life", jointly sponsored by the People's Government of Guangzhou Municipality, the Bureau of Civil Affairs of Guangzhou Municipality, and the Zhongshan Ophthalmic Center (ZOC), has been initiated in Guangzhou to implement a program of free clinics in parks and free cataract surgery targeting the impoverished population living in urban China in 2012. After 3 years' exploration, the management mode of this program has been perfected, and approximately 4000 cataract surgeries had been performed on the low-income elderly.

Although there are a large number of poor communities throughout the country, free cataract surgery programs in poor urban China are restricted to several metropolises due to limited medical resources and social overlook. Fully understanding patient satisfaction regarding the free cataract surgery program and understanding the patient characteristics of this special, neglected community may contribute to the improvement and the further expansion of the management mode of free cataract surgery programs.

DETAILED DESCRIPTION:
Age-related cataracts remain the leading cause of treatable blindness in China. The prevalence of cataract blindness continues to climb due to the expanding elderly subpopulation. Surgery is the only available treatment; however, the cataract surgical rate (CSR) in China remains relatively low (772 cases per million per year) relative to affluent countries (6000 cases per million per year) or certain developing areas (2672 cases per million per year). Studies have reported that the primary barrier to cataract surgery is financial difficulty, and this challenge could be efficiently addressed by reducing the surgical fee1 or providing free cataract surgery. However, the prices, availability and affordability of medicines or medical services to the poor in China require further improvement, according to the standards developed by the World Health Organization (WHO) in collaboration with Health Action International (HAI) in May 2003. Although a host of free cataract screening and surgery programs have been widely implemented in rural areas of China in conjunction with a new national healthcare reform officially launched in 2009 to tackle high medical expenses, including promoting free medical treatments, free cataract surgery programs have rarely been implemented in financially-challenged urban China. Even in Guangzhou, one of the largest metropolises in China, many low-income cataract patients, a neglected cohort, continue to need cataract surgery. A program titled "care for your eyes, lighten your life", jointly sponsored by the People's Government of Guangzhou Municipality, the Bureau of Civil Affairs of Guangzhou Municipality, and the Zhongshan Ophthalmic Center (ZOC), has been initiated in Guangzhou to implement a program of free clinics in parks and free cataract surgery targeting the impoverished population living in urban China in 2012.13 After 3 years' exploration, the management mode of this program has been perfected, and approximately 4000 cataract surgeries had been performed on the low-income elderly.

Although there are a large number of poor communities throughout the country, free cataract surgery programs in poor urban China are restricted to several metropolises due to limited medical resources and social overlook. Fully understanding patient satisfaction regarding the free cataract surgery program and understanding the patient characteristics of this special, neglected community may contribute to the improvement and the further expansion of the management mode of free cataract surgery programs. In this telephone survey, the investigators aimed to investigate the characteristics of the low-income patients undergoing free cataract surgery, including patient demographics, patient resource, health conditions, reasons for choosing the free surgery, and overall evaluation of the free cataract surgery program.

ELIGIBILITY:
Inclusion Criteria:

* All participants with presenting visual acuity (PVA), unaided visual acuity or aided visual acuity with walk-in optical correction5 of ≤20/50 in either eye.

Exclusion Criteria:

* Patients with severe eye diseases and bad general condition were excluded.

Ages: 50 Years to 102 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: A free cataract surgery program was jointly initiated by the People's Government of Guangzhou Municipality, the Bureau of Civil Affairs of Guangzhou Municipality, and the ZOC in May 2012. Guangzhou citizens aged ≥50 years with low income who relied on social subsidies were candidates for this activity.
Sampling Method: Probability Sample
Enrollment: 883 (Actual)
Dates: Start 2012-05; Primary Completion 2014-08 (Actual); Study Completion 2014-08 (Actual)

PRIMARY OUTCOMES:
Family income of the low-income elderly who underwent free cataract surgery assessed through telephone survey | 9 months after surgery

SECONDARY OUTCOMES:
the education level of the low-income elderly who underwent free cataract surgery through telephone survey | 9 months after surgery

CONTACTS AND LOCATIONS:
Overall Officials: Weirong Chen, M.D., Study Director — Zhongshan Ophthalmic Center, Sun Yat-sen University; Yizhi Liu, M.D.;Ph.D., Study Chair — Zhongshan Ophthalmic Center, Sun Yat-sen University; Haotian Lin, M.D.;Ph.D., Principal Investigator — Zhongshan Ophthalmic Center, Sun Yat-sen University
Locations (1):
- Zhognshan Ophthalmic Center, Sun Yat-sen University, Guangzhou, Guangdong, China

REFERENCES:
- [Background] Vision 2020: the cataract challenge. Community Eye Health. 2000;13(34):17-9. No abstract available. PMID 17491949
- [Background] Wang Y, Wang J, Maitland E, Zhao Y, Nicholas S, Lu M. Growing old before growing rich: inequality in health service utilization among the mid-aged and elderly in Gansu and Zhejiang Provinces, China. BMC Health Serv Res. 2012 Sep 4;12:302. doi: 10.1186/1472-6963-12-302. PMID 22947369
- [Background] Liang YB, Friedman DS, Wong TY, Zhan SY, Sun LP, Wang JJ, Duan XR, Yang XH, Wang FH, Zhou Q, Wang NL; Handan Eye Study Group. Prevalence and causes of low vision and blindness in a rural chinese adult population: the Handan Eye Study. Ophthalmology. 2008 Nov;115(11):1965-72. doi: 10.1016/j.ophtha.2008.05.030. Epub 2008 Aug 5. PMID 18684506
- [Background] Xu J, Zhu S, Li S, Pizzarello L. Models for improving cataract surgical rates in southern China. Br J Ophthalmol. 2002 Jul;86(7):723-4. doi: 10.1136/bjo.86.7.723. PMID 12084736
- [Background] Zhang XJ, Liang YB, Liu YP, Jhanji V, Musch DC, Peng Y, Zheng CR, Zhang HX, Chen P, Tang X, Lam DS. Implementation of a free cataract surgery program in rural China: a community-based randomized interventional study. Ophthalmology. 2013 Feb;120(2):260-5. doi: 10.1016/j.ophtha.2012.07.087. Epub 2012 Oct 27. PMID 23107580
- [Derived] Lin H, Lin D, Long E, Jiang H, Qu B, Tang J, Lin Y, Chen J, Wu X, Lin Z, Li X, Liu Z, Zhang B, Chen H, Tan X, Luo L, Liu Y, Chen W. Patient participation in free cataract surgery: a cross-sectional study of the low-income elderly in urban China. BMJ Open. 2016 Apr 15;6(4):e011061. doi: 10.1136/bmjopen-2016-011061. PMID 27084286
- See also: Home page of Zhongshan Ophthalmic Center — http://www.gzzoc.com/